CLINICAL TRIAL: NCT04435457
Title: Uncovering the Cardiac Phenotype of Individuals With SARS-COV-2 and Cardiac Injury
Brief Title: Cardiovascular Implications of COVID-19
Status: Terminated | Type: Observational
Why Stopped: COVID-19 natural history has changed and no further patients meet eligibility as hospitalizations are at a minimum.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Justin Grodin, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0359
Record Dates: First submitted 2020-06-02; First posted 2020-06-17 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV 2; SARS Pneumonia; COVID-19; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere; Cardiac Complication
Keywords: SARS-CoV 2; Troponin; Cardiac injury; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — A fasting venous blood sample (50 cc) will be collected, maintained on ice and transported to the Mammen Laboratory, which is located on the campus of UT Southwestern. Both serum and plasma will be isolated and aliquoted for storage and immediately frozen and stored until use and will not undergo any freeze-thaw cycles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At the end of December of 2019, a series of patients in Wuhan, China were struck with a mysterious respiratory infection. These isolated events have rapidly grown into a deadly, global pandemic. This pandemic is caused by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), which results in the Coronavirus Disease 2019 (COVID-19). For individuals infected with COVID-19, approximately 30% of the hospitalized cases are associated with cardiovascular complications. Data are emerging that individuals with pre-exiting conditions (like hypertension, diabetes, cancer, or medical issues related to the immune system) are most susceptible to complications related to COVID-19. Furthermore, individuals of certain racial and ethnic backgrounds (e.g. African American and Hispanic) are at a higher risk of death from COVID-19. Despite these emerging observations, it remains unclear who will develop the cardiovascular complications (acute myocardial injury with evidence of a myocarditis-like picture and cardiogenic shock) and what the long term sequelae of this disease will be for survivors of this infection after hospitalization. Thus, the goals of this project are to better understand the epidemiology of cardiac injury in acutely ill COVID-19 patients through deep cardiac phenotyping and identify the molecular profile of individuals most susceptible to cardiac injury from COVID-19.

DETAILED DESCRIPTION:
This will be a cross-sectional cohort study of participants who will undergo a detailed cardiovascular imaging evaluation and blood draw once they have recuperated from a prior index-hospitalization at Clements University Hospital or Parkland Memorial Hospital in Dallas, Texas, USA for COVID-19 and are no longer contagious (~4-6 weeks post hospitalization). Due to the uncertainty with which the extent of cardiac injury represents phenotypic cardiac manifestations in COVID-19, the investigators plan to enroll individuals according to their highest, in-hospital, (high sensitivity - cardiac troponin T) hs-cTnT. The following proposed stratification scheme will afford testing a spectrum hs-cTnT levels.

Table: Enrollment strata by hs-cTnT (N=70)

hs-cTnT [ng/L] < 50 50-100 101-500 > 500

Enrollment N=20 N=20 N=20 N=10

The investigators propose the following exploratory protocol for deep phenotyping to characterize surviving patients with COVID-19 and elevated hs-cTnT during hospitalization.

All participants will undergo a protocolized multiparametric cardiac magnetic resonance imaging (CMR) assessment with an electrocardiography-gated breath hold protocol under the oversight of study personnel and read by a reader blinded to hs-cTnT data from the COVID-19 index hospitalization. Conventional 1H CMR evaluations will include T2 maps, native and post-contrast T1 maps, as well as extracellular volume index calculation and late gadolinium for inflammatory injury. Standardized adenosine hyperemic stress perfusion CMR will be performed for quantitative myocardial blood flow analysis. In addition to conventional 1H CMR a subset of 5 patients from the highest and lowest troponin groups, age- and BMI-matched, will undergo hyperpolarized 13C metabolic CMR with infusion of [1-13C] pyruvate under fasting conditions to assess inflammation and post carbohydrate load to assess a decrease in myocardial mitochondrial oxidative metabolism.

Biospecimens will be collected by study personnel at the time of CMR or preliminary study site visit. A fasting venous blood sample (50 cc) will be collected, maintained on ice and transported to the Mammen Laboratory, which is located on the campus of UT Southwestern. Both serum and plasma will be isolated and aliquoted for storage and immediately frozen and stored until use and will not undergo any freeze-thaw cycles. RNA and protein will be extracted from the samples for biomarker and autoantibody (AAb) assays. The presence of cardiac-specific AAbs has been shown to be involved in both the manifestation and development of cardiac disease manifestation and predicting disease development. Utilizing a customized ELISA-based detection assay, ~20 circulating cardiac-specific AAbs that have been reported to be associated with heart failure will be assessed and quantified during the early (1-2 months post-hospitalization) phases of the patient post COVID-19 hospitalization course.

Leukocytes will be isolated from the biospecimens samples and genomic DNA will be extracted from the cells to perform Next Generation Whole Exome Sequencing (WES). These studies will be undertaken in the Next-Generation Sequencing Core on campus. Capitalizing on a well-established research collaboration between the Mammen Laboratory and the McDermott bioinformatics group, the WES data will be analyzed for genetic mutations associated with cardiomyopathy as well as autoimmunity.

If funds are available, both the imaging and molecular assessments will be duplicated in individuals with paired data after an additional 10-12 months from hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women 18-80 years old who were previously hospitalized with confirmed COVID-19
* Were alive at the time of discharge from COVID-19 hospitalization
* Had measured hs-cTnT levels during hospitalization

Exclusion Criteria:

* Prior cardiovascular disease (before COVID-19 infection), defined as self-reported history or electronic medical record diagnosis of cardiac arrest, myocardial infarction, coronary revascularization, heart failure, or stroke prior to COVID-19 hospitalization
* Urgent-coronary revascularization or type I myocardial infarction within the preceding 30 days
* Cardiac transplantation
* Body weight >250 lbs
* Moderate to severe chronic renal dysfunction defined by an eGFR ≤30 mL/min/1.73 m2
* Inability to safely undergo a CMR
* Unwilling or unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adults with a prior hospitalization for COVID-19 at either Parkland Memorial Hospital or Clements University Hospital in Dallas, Texas, USA who have recovered and are no-longer at-risk of COVID-19 disease transmission according the United States Centers for Disease Control guidelines will be considered for inclusion.
  All patients admitted to either hospital with suspected or confirmed COVID-19 receive an in-hospital standard-of-care metabolic, cardiac, and inflammatory biomarker protocolized assessment that includes daily basic metabolic panels, complete blood counts with differential, hs-cTnT, and C-reactive protein (CRP) coupled with every third day amino terminal pro-B-type natriuretic peptide (NT-proBNP), D-dimer, and ferritin. These labs are obtained from the day of admission to discharge. ]
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Myocarditis | Up to 4 weeks
  Patterns of late gadolinium enhancement and T1 and T2 mapping consistent with myocarditis on a post-hospitalization cardiac magnetic resonance imaging examination

SECONDARY OUTCOMES:
Prevalence of cardiac abnormalities by cardiac magnetic resonance imaging | Up to 4 weeks
  This includes categorically abnormal structural, mechanical functional, vascular, and metabolic using cardiac magnetic resonance imaging
Prevalence of molecular and genetic immune system abnormalities | Up to 4 weeks
  Presence of cardiac autoantibodies and defects within the immune system as detected by Whole Exome Sequencing making an individual susceptible to subacute cardiac injury during COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Grodin, MD, MPH, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided